CLINICAL TRIAL: NCT00996996
Title: Phase II Trial of Iodine-131 Anti-B1 Antibody for Previously Untreated, Advanced Stage, Low Grade Non-Hodgkin's Lymphoma
Brief Title: Iodine-131 Anti-B1 Antibody (Tositumomab and Iodine I 131 Tositumomab) for Previously Untreated, Advanced-stage, Low Grade Non-Hodgkin's Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 104517
Record Dates: First submitted 2009-10-08; First posted 2009-10-16 (Estimated); Results first posted 2012-07-04 (Estimated); Last update posted 2017-01-11 (Estimated); Status verified 2016-11

CONDITIONS: Lymphoma, Non-Hodgkin
Keywords: Radioimmunotherapy; Anti-B1 Antibody and Iodine-131 Anti-B1 Antibody; Tositumomab and Iodine I 131 Tositumomab; non-Hodgkin's Lymphoma; Bexxar
MeSH Terms: conditions — Lymphoma, Non-Hodgkin | interventions — tositumomab I-131

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- open-label, single arm (Experimental): Tositumomab and Iodine I 131 Tositumomab
  Interventions: Biological: Tositumomab and Iodine I 131 Tositumomab (Anti-B1 Antibody and Iodine-131 Anti-B1 Antibody)

INTERVENTIONS:
Biological: Tositumomab and Iodine I 131 Tositumomab (Anti-B1 Antibody and Iodine-131 Anti-B1 Antibody) — Dosimetric Dose: 450 mg of Anti-B1 Antibody infused over 70 minutes (inclusive of a 10-minute flush) immediately followed by 5 mCi (35 mg) of Iodine-131 Anti-B1 Antibody infused over 30 minutes (inclusive of a 10-minute flush).
  Therapeutic Dose: Seven to 14 days after the dosimetric dose, 450 mg of Anti-B1 Antibody infused over 70 minutes (inclusive of a 10-minute flush), immediately followed by the patient-specific milliCurie activity (35 mg) of Iodine-131 Anti-B1 Antibody to deliver a total body dose (TBD) of 75 cGy infused over 30 minutes (inclusive of a 10-minute flush). Obese patients were dosed based upon 137% of their calculated lean body mass.

SUMMARY:
This is a single-arm, single-institution, phase II study of Iodine-131 Anti-B1 Antibody for patients with previously untreated, advanced-stage (stage III or IV) low-grade non-Hodgkin's B-cell lymphoma. A total of 75-80 patients will be enrolled.

Patients will undergo two phases of the study. In the first phase, termed the "dosimetric dose", patients will receive an infusion of unlabeled Anti-B1 Antibody (450 mg) over 70 minutes (including a 10-minute flush) immediately followed by a 30-minute infusion (including a 10-minute flush) of Anti-B1 Antibody (35 mg) which has been trace-labeled with 5 mCi of Iodine-131. Whole body gamma camera scans will be obtained 5 to 8 times between Days 0 and 7 following the dosimetric dose. Using the dosimetric data from 3 imaging timepoints (the imaging timepoints to be used in decreasing order of preference depending on availability of data are Days 0, 3, and 7; Days 0, 4, and 7; Days 0, 3 and 6; Days 0, 4, and 6; Days 0, 2, and 7; and Days 0, 2, and 6), a patient-specific dose of Iodine- 131 to deliver the desired total body dose of radiotherapy will be calculated. In the second phase, termed the "therapeutic dose", patients will receive a 70-minute infusion (including a 10-minute flush) of unlabeled Anti-B1 Antibody (450 mg) immediately followed by a 30-minute infusion (including a 10-minute flush) of Anti-B1 Antibody (35 mg) labeled with the patient-specific dose of Iodine-131 to deliver a whole body dose of 75 cGy. Patients who are obese will be dosed based upon 137% of their calculated lean body mass. Patients will be treated with either saturated solution potassium iodide (SSKI), Lugol's solution, or potassium iodide tablets starting at least 24 hours prior to the first infusion of the Iodine-131 Anti-B1 Antibody (i.e., dosimetric dose) and continuing for 14 days following the last infusion of Iodine-131 Anti-B1 Antibody (i.e., therapeutic dose).

The primary endpoint of the study is the determination of the response rate with Iodine-131 Anti-B1 Antibody in previously untreated patients with low-grade non-Hodgkin's lymphoma (NHL). The secondary endpoints include duration of response, safety, radiation dosimetry, and the predictive value of detection of the presence or absence minimal residual disease by molecular techniques on response duration.

ELIGIBILITY:
Inclusion Criteria

* Patients must have a histologically confirmed diagnosis of lowgrade non-Hodgkin's B-cell lymphoma. The following low-grade histologies are included: small lymphocytic (with or without plasmacytoid differentiation); follicular, small cleaved; follicular, mixed small cleaved and follicular large cell (less than 50% large cell component); and monocytoid B-cell lymphoma.
* Patients must have evidence that their tumor tissue expresses the CD20 antigen. Immunoperoxidase stains of paraffin-embedded tissue showing positive reactivity with L26 antibody or immunoperoxidase stains of frozen tissue showing positive reactivity with Anti-B1 Antibody (Coulter Clone®) or similar commercially available CD20 antibody (>50% of tumor cells are positive) or evidence of CD20 positivity by flow cytometry (>50% of tumor cells are positive) are acceptable evidence of CD20 positivity. Testing of tumor tissue from any time in the course of the patient's disease is acceptable.
* Patients must have Ann Arbor stage III or IV extent of disease after complete staging.
* Patients must not have had any previous treatment for low-grade lymphoma including chemotherapy or radiation. They may be newly diagnosed or observed without treatment after diagnosis. Symptomatic and asymptomatic patients will be eligible.
* Patients must have a performance status of at least 60% on the Karnofsky Scale and an anticipated survival of at least 3 months.
* Patients must have an absolute neutrophil count (ANC) >1500 cells/mm3 and a platelet count >100,000 cells/mm3 within 14 days of study entry. These blood counts must be sustained without support of hematopoietic cytokines or transfusion of blood products.
* Patients must have adequate renal function (defined as serum creatinine <1.5 x upper limit of normal [ULN]) and hepatic function (defined as total bilirubin <1.5 x ULN and aspartate transaminase [AST] <5 x ULN) within 14 days of study entry.
* Patients must have bi-dimensionally measurable disease. At least one lesion must be ≥2 x 2 cm (by computed tomography [CT] scan).
* Patients must be at least 18 years of age.
* Patients must give written informed consent and sign an IRB- approved informed consent form prior to study entry.

Exclusion Criteria

* Patients with more than an average of 25% of the intratrabecular marrow space involved by lymphoma in bone marrow biopsy specimens as assessed microscopically within 42 days of study entry. Bilateral posterior iliac crest core biopsies are required if the percentage of intratrabecular space involved exceeds 10% on a unilateral biopsy. The mean of bilateral biopsies must be no more than 25%.
* Patients with evidence of active infection requiring intravenous (IV) antibiotics at the time of study entry.
* Patients with New York Heart Association class III or IV heart disease or other serious illness that would preclude evaluation.
* Patients with active obstructive hydronephrosis.
* Patients with prior malignancy other than lymphoma, except for adequately treated skin cancer, in situ cervical cancer, or other cancer for which the patient has been disease-free for 5 years.
* Patients with known HIV infection.
* Patients with known brain or leptomeningeal metastases.
* Patients who are pregnant or nursing. Patients of childbearing potential must undergo a pregnancy test within 7 days of study entry and radiolabeled antibody is not to be administered until a negative result is obtained. Males and females must agree to use effective contraception for 6 months following the radioimmunotherapy.
* Patients with previous allergic reactions to iodine. This does not include reacting to IV iodine-containing contrast materials.
* Patients who were previously given any monoclonal or polyclonal antibodies of any non-human species for either diagnostic or therapeutic purposes. This includes engineered chimeric and humanized antibodies.
* Patients who are concurrently receiving either approved or nonapproved (through another protocol) anti-cancer drugs or biologics.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 77 (Actual)
Dates: Start 1996-06; Primary Completion 1999-03 (Actual); Study Completion 2011-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Individual Participant Data Set: 104517 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 104517 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 104517 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 104517 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 104517 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 104517 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 104517 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Groups:
- Tositumomab and Iodine I-131 Tositumomab: Dosimetric dose (administered only once on Day 0): 450 milligrams (mg) unlabeled tositumomab administered intravenously (IV) over 70 minutes, followed immediately by 5 millicurie (mCi) iodine I-131 tositumomab (contained in 35 mg tositumomab) infused over 30 minutes. Therapeutic dose (administered only once 7 to 14 days after the dosimetric dose): 450 mg unlabeled tositumomab administered IV over 70 minutes, followed immediately by iodine I-131 tositumomab (contained in 35 mg tositumomab) administered IV infused over 30 minutes. The dose was calculated based on the dosimetric dose results to deliver a total body radiation dose of 75 centigray (cGy).
Period: Overall Study
Arm/Group | Tositumomab and Iodine I-131 Tositumomab
Started | 77
Completed | 44 (These participants completed 12 years of follow-up.)
Not Completed | 33
Not completed — Progressive Disease | 10
Not completed — Non-compliance | 8
Not completed — Lost to Follow-up | 9
Not completed — Death | 5
Not completed — Did Not Receive Study Medications | 1

BASELINE CHARACTERISTICS:
Arm/Group | Tositumomab and Iodine I-131 Tositumomab
Number analyzed (Participants) | 76
Age, Continuous [Mean (Standard Deviation); unit: Years] — Baseline characteristics are summarized for the Intent-to-Treat (ITT)-Exposed Population, comprised of all participants who were enrolled in the study and received at least one dose of study drug. A total of 77 participants were enrolled in the study; however, only 76 participants received study drug.
  Years | 48.1 (9.9)
Gender [Count of Participants; unit: Participants] — Baseline characteristics are summarized for the ITT-Exposed Population, comprised of all participants who were enrolled in the study and received at least one dose of study drug. A total of 77 participants were enrolled in the study; however, only 76 participants received study drug.
  Participants
    Female | 35
    Male | 41
Race/Ethnicity, Customized [Number; unit: participants] — Baseline characteristics are summarized for the ITT-Exposed Population, comprised of all participants who were enrolled in the study and received at least one dose of study drug. A total of 77 participants were enrolled in the study; however, only 76 participants received study drug.
  participants
    White | 74
    Hispanic | 1
    Asian | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Confirmed Response, Including Participants With Complete Response (CR), Clinical Complete Response (CCR), and Partial Response (PR)
Description: Confirmed response required CR, CCR, or PR, which were confirmed by 2 separate response evaluations >=4 weeks apart. CR: Complete resolution of all disease-related radiological abnormalities and disappearance of all signs and symptoms related to the disease. CCR: Complete resolution of all disease-related symptoms, but residual foci, thought to be residual scar tissue, are present. PR: >=50% reduction in the sum of the products of the longest perpendicular diameters of all measurable lesions with no new lesions.
Time Frame: From Study Day 0 (start of treatment) up to 12 years (long-term follow up)
Population: ITT-Exposed Population: all participants who were enrolled in the study and received at least one dose of study drug. Only participants evaluable for confirmed response were assessed.
Measure: Number; unit: participants
Arm/Group | Tositumomab and Iodine I-131 Tositumomab
Number analyzed (Participants) | 75
participants | 72
Statistical Analysis 1: Comparison: Tositumomab and Iodine I-131 Tositumomab; Test type: Superiority or Other; Percentage of participants = 95, 95% CI 2-sided [90 to 100] — The estimated value represents the percentage of participants with a confirmed response

2. Primary Outcome: Number of Participants With Response, Including Participants With Complete Response (CR), Clinical Complete Response (CCR), or Partial Response (PR)
Description: CR: Complete resolution of all disease-related radiological abnormalities and disappearance of all signs and symptoms related to the disease. CCR: Complete resolution of all disease-related symptoms, but residual foci, thought to be residual scar tissue, are present. PR: >=50% reduction in the sum of the products of the longest perpendicular diameters of all measurable lesions with no new lesions.
Time Frame: From Study Day 0 (start of treatment) up to 12 years (long-term follow up)
Population: ITT-Exposed Population
Measure: Number; unit: participants
Arm/Group | Tositumomab and Iodine I-131 Tositumomab
Number analyzed (Participants) | 76
participants | 74
Statistical Analysis 1: Comparison: Tositumomab and Iodine I-131 Tositumomab; Test type: Superiority or Other; Percentage of participants = 97, 95% CI 2-sided [94 to 100] — The estimated value represents the percentage of participants with a response

3. Primary Outcome: Number of Participants With Confirmed Complete Response (CR, CCR, and CR+CCR) and Partial Response (PR)
Description: Responses were confirmed by two separate response evaluations at least 4 weeks apart. CR: Complete resolution of all disease-related radiological abnormalities and disappearance of all signs and symptoms related to the disease. CCR: Complete resolution of all disease-related symptoms, but residual foci, thought to be residual scar tissue, are present. PR: >=50% reduction in the sum of the products of the longest perpendicular diameters of all measurable lesions with no new lesions.
Time Frame: From Study Day 0 (start of treatment) up to 12 years (long-term follow up)
Population: ITT-Exposed Population. Only participants evaluable for confirmed response (R) were assessed. R had to be confirmed by a consecutive R that was the same or better >=4 weeks apart. Each individual confirmed R category only counts the R confirmed by the exact same R; therefore, not all possible combinations are represented in the table.
Measure: Number; unit: participants
Arm/Group | Tositumomab and Iodine I-131 Tositumomab
Number analyzed (Participants) | 75
participants
  CR | 53
  CCR | 2
  CR+CCR | 57
  PR | 13
Statistical Analysis 1: Comparison: Tositumomab and Iodine I-131 Tositumomab; Test type: Superiority or Other; Percentage of participants = 70, 95% CI 2-sided [59 to 80] — The estimated value represents the percentage of participants with a confirmed CR
Statistical Analysis 2: Comparison: Tositumomab and Iodine I-131 Tositumomab; Test type: Superiority or Other; Percentage of participants = 3, 95% CI 2-sided [0 to 6] — The estimated value represents the percentage of participants with a confirmed CCR
Statistical Analysis 3: Comparison: Tositumomab and Iodine I-131 Tositumomab; Test type: Superiority or Other; Percentage of participants = 75, 95% CI 2-sided [65 to 85] — The estimated value represents the percentage of participants with confirmed CR + confirmed CCR
Statistical Analysis 4: Comparison: Tositumomab and Iodine I-131 Tositumomab; Test type: Superiority or Other; Percentage of participants = 17, 95% CI 2-sided [9 to 26] — The estimated value represents the percentage of participants with a confirmed PR

4. Primary Outcome: Number of Participants With Complete Response (CR, CCR, and CR+CCR) and Partial Response (PR)
Description: as for outcome 2
Time Frame: From Study Day 0 (start of treatment) up to 12 years (long-term follow up)
Population: ITT-Exposed Population
Measure: Number; unit: participants
Arm/Group | Tositumomab and Iodine I-131 Tositumomab
Number analyzed (Participants) | 76
participants
  CR | 56
  CCR | 3
  CR+CCR | 59
  PR | 15
Statistical Analysis 1: Comparison: Tositumomab and Iodine I-131 Tositumomab; Test type: Superiority or Other; Percentage of participants = 74, 95% CI 2-sided [64 to 84] — The estimated value represents the percentage of participants with a CR
Statistical Analysis 2: Comparison: Tositumomab and Iodine I-131 Tositumomab; Test type: Superiority or Other; Percentage of participants = 4, 95% CI 2-sided [0 to 8] — The estimated value represents the percentage of participants with a CCR
Statistical Analysis 3: Comparison: Tositumomab and Iodine I-131 Tositumomab; Test type: Superiority or Other; Percentage of participants = 78, 95% CI 2-sided [68 to 87] — The estimated value represents the percentage of participants with a CR + CCR
Statistical Analysis 4: Comparison: Tositumomab and Iodine I-131 Tositumomab; Test type: Superiority or Other; Percentage of participants = 20, 95% CI 2-sided [11 to 29] — The estimated value represents the percentage of participants with a PR

5. Secondary Outcome: The Estimated Value Represents the Percentage of Participants With a PR
Description: Duration of response (CR, CCR, or PR) is defined as the time from the first documented response to the first documented progression. Progressive Disease (PD) is defined as a >=25% increase from the nadir value of the sum of the products of the longest perpendicular diameters of all measurable lesions or the appearance of any new lesion.
Time Frame: From Study Day 0 (start of treatment) up to 12 years (long-term follow up)
Population: ITT-Exposed Population. Only participants who experienced confirmed CR, CCR, or PR with PD were assessed. Response (R) had to be confirmed by a consecutive R that was the same or better >=4 weeks apart. Each individual confirmed R category only counts the R confirmed by the exact same R; therefore, not all possible combinations are represented.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Tositumomab and Iodine I-131 Tositumomab
Number analyzed (Participants) | 45
months
  Confirmed CR+CCR+PR, n=45 | 98.0 [34.5 to 130.7]
  Confirmed CR+CCR, n=30 | 129.2 [98.3 to NA] — The SAS procedure was not able to calculate the upper limit of the confidence interval because there were too few events.
  Confirmed PR, n=13 | 6.9 [5.2 to 8.8]
  Confirmed CR, n=27 | 130.7 [106.4 to NA] — The SAS procedure was not able to calculate the upper limit of the confidence interval because there were too few events.
  Confirmed CCR, n=2 | 11.8 [4.7 to 18.9]

6. Secondary Outcome: Overall Survival
Description: Overall survival is defined as the time from the treatment start date to the date of death from any cause.
Time Frame: From Study Day 0 (start of treatment) up to 12 years (long-term follow up)
Population: ITT-Exposed Population. Only those participants who died during the study due to any cause were assessed.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Tositumomab and Iodine I-131 Tositumomab
Number analyzed (Participants) | 15
months | NA [NA to NA] — The SAS procedure was not able to calculate the median or the confidence interval because there were too few events.

7. Secondary Outcome: Time to Progression of Disease or Death (Progression-free Survival)
Description: Time to progression is defined as the time from the treatment start date to the first documented progression or death. Progressive Disease is defined as a >=25% increase from the nadir value of the sum of the products of the longest perpendicular diameters of all measurable lesions or the appearance of any new lesion.
Time Frame: From Study Day 0 (start of treatment) up to 12 years (long-term follow up)
Population: ITT-Exposed Population. Only those participants who experienced disease progression or died were assessed.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Tositumomab and Iodine I-131 Tositumomab
Number analyzed (Participants) | 51
months | 74.3 [32.4 to 118.2]

8. Secondary Outcome: Number of Participants With Resolution of All Baseline B-symptoms by the End of the Study
Description: The Ann Arbor staging system of lymphomas is used to summarize the extent of the cancer's spread. Stages are classified by Roman numerals I (less spread) to IV (more spread). If the following symptoms (called B-symptoms) are present, a "B" classification is added to the stage: night sweats, intermittant fever, and weight loss. B-symptoms indicate the presence of systemic symptoms. The presence or absence of B-symptoms has prognostic significance and is reflected in the staging of these lymphomas.
Time Frame: Baseline and up to 12 years (long-term follow up)
Population: ITT-Exposed Population. Only those participants who experienced any B-symptom at Baseline were assessed. Not all participants experienced all B-symptoms at Baseline; thus, the number of participants analyzed represents all participants who experienced at least one B-symptom.
Measure: Number; unit: participants
Arm/Group | Tositumomab and Iodine I-131 Tositumomab
Number analyzed (Participants) | 11
participants
  Night sweats, n=8 | 8
  Intermittant fever, n=3 | 3
  Weight loss, n=4 | 4

9. Secondary Outcome: Number of Participants Who Were Polymerase Chain Reaction (PCR)-Positive at Baseline With Bone Marrow Conversion to a Status of PCR Positive and Negative Any Time After Treatment
Description: PCR is a scientific technique in molecular biology to amplify a single copy or a few copies of a piece of deoxyribonucleic acid (DNA) across several orders of magnitude, generating thousands to millions of copies of a particular DNA sequence. Applications of PCR technique include: selective DNA isolation, amplification and quantification of DNA, and the diagnosis of diseases. PCR positive: interchromosomal translocation t(14;18) is present. PCR negative: t(14;18) is absent.
Time Frame: Baseline and up to 12 years (long-term follow up)
Population: ITT-Exposed Population. Only those participants with a PCR-positive status at Baseline were assessed. One participant had a Baseline measurement but no post Baseline measure, and was thus not assessed.
Measure: Number; unit: participants
Arm/Group | Tositumomab and Iodine I-131 Tositumomab
Number analyzed (Participants) | 40
participants
  PCR Positive after treatment | 1
  PCR Negative after treatment | 38

10. Secondary Outcome: Duration of Response (the Time From the First Documented Response to the First Documented Progression) for Participants Who Were PCR Positive at Baseline and Converted to PCR Negative Status After Treatment
Description: as for outcome 9
Time Frame: Baseline and up to 12 years (long-term follow up)
Population: ITT-Exposed Population. Only those participants who were PCR positive at Baseline and converted to a status of PCR negative were assessed.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Tositumomab and Iodine I-131 Tositumomab
Number analyzed (Participants) | 38
months
  All responders (CR+CCR+PR), n=38 | 59.5 [26.9 to 106.4]
  Complete responders (CR+CCR), n=30 | 98.2 [35.5 to NA] — The SAS procedure was not able to calculate the confidence interval because there were too few events.
  Partial responders, n=8 | 6.9 [4.4 to 10.6]

11. Secondary Outcome: Progression-free Survival (PFS) Based on Participants' Baseline PCR Status
Description: PCR is a scientific technique in molecular biology to amplify a single copy or a few copies of a piece of deoxyribonucleic acid (DNA) across several orders of magnitude, generating thousands to millions of copies of a particular DNA sequence. Applications of PCR technique include: selective DNA isolation, amplification and quantification of DNA, and the diagnosis of diseases. PCR positive: interchromosomal translocation t(14;18) is present. PCR negative: t(14;18) is absent. PFS is defined as the time from the dosimetric dose to the first documented occurrence of disease progression or death.
Time Frame: Baseline and up to 12 years (long-term follow up)
Population: ITT-Exposed Population. Only those participants with a PCR status taken at Baseline were evaluated for PFS.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Tositumomab and Iodine I-131 Tositumomab
Number analyzed (Participants) | 73
months
  PCR-negative participants, n=33 | 130.8 [70.3 to NA] — The SAS procedure was not able to calculate the upper limit of the confidence interval because there were too few events.
  PCR-positive participants, n=40 | 48.8 [20.7 to 100.0]

12. Secondary Outcome: Initial Half-life (t1/2alpha)
Description: t1/2 alpha is the estimated initial or alpha phase half-life in a two-compartmental pharmacokinetic model. Half-life measures how long it takes for the concentration of drug in the blood to decrease by half.
Time Frame: 0-120 hours from the dosimetric dose (given only on Day 0) and 0-120 hours from the therapeutic dose (given only on Day 7)
Population: ITT-Exposed Population. Only those participants for whom pharmacokinetic blood samples were collected at the indicated time points were assessed.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Tositumomab and Iodine I-131 Tositumomab
Number analyzed (Participants) | 68
hours | 3.85 (3.33)

13. Secondary Outcome: Terminal Half-life (t1/2beta)
Description: t1/2 beta is the estimated terminal or beta phase half-life in a two-compartmental pharmacokinetic model. Half-life measures how long it takes for the concentration of drug in the blood to decrease by half.
Time Frame: as for outcome 12
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Tositumomab and Iodine I-131 Tositumomab
Number analyzed (Participants) | 70
hours | 64.57 (16.23)

14. Secondary Outcome: Area Under the Curve (AUC) at 0 to 120 Hours and 0 to Infinity Hours
Description: Area under the concentration-time curve for I-131 tositumomab from time 0 to 120 hours and time 0 to infinity hours (extrapolated) after the end of the dosimetric dose infusion was measured. Unit: %ID*h/ml, where %ID/ml is the percentage of the injected dose per milliliter of blood. AUC measures how much drug is in the system over time after infusion.
Time Frame: 0-120 hours and 0-infinity hours from the dosimetric dose (given only on Day 0) and 0-120 hours and 0-infinity hours from the therapeutic dose (given only on Day 7)
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: %ID*h/ml
Arm/Group | Tositumomab and Iodine I-131 Tositumomab
Number analyzed (Participants) | 70
%ID*h/ml
  AUC(0-infinity) | 1.43 (0.41)
  AUC(0-120) | 1.03 (0.26)

15. Secondary Outcome: Clearance Values
Description: Clearance of I-131 tositumomab after intravenous administration was measured. The clearance of a drug measures the rate at which the drug is removed from the body after the dose.
Time Frame: as for outcome 12
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: Milliliters per hour (ml/hr)
Arm/Group | Tositumomab and Iodine I-131 Tositumomab
Number analyzed (Participants) | 70
Milliliters per hour (ml/hr) | 77.34 (28.73)

16. Secondary Outcome: Maximum Concentration (Cmax) Values
Description: Cmax is the maximum observed I-131 tositumomab concentration from time zero (end of the dosimetric dose infusion) to 120 hours after the end of the infusion. Unit: %ID/ml, where %ID/ml is the percentage of the injected dose per milliliter of blood. Cmax is the highest drug concentration in the blood after infusion.
Time Frame: as for outcome 12
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: %ID/ml
Arm/Group | Tositumomab and Iodine I-131 Tositumomab
Number analyzed (Participants) | 70
%ID/ml | 0.020 (0.005)

17. Secondary Outcome: Volume of Distribution at Infusion Time 0 (Vd0) and Steady State (Vdss)
Description: Volume of distribution at the start of infusion and at steady state of I-131 tositumomab. The volume of distribution measures how much the drug spreads through the body after the dose. Steady state is defined as that state at which the overall intake of a drug is fairly in dynamic equilibrium with its elimination.
Time Frame: as for outcome 12
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: milliliters (ml)
Arm/Group | Tositumomab and Iodine I-131 Tositumomab
Number analyzed (Participants) | 70
milliliters (ml)
  Vd0 | 5297 (1123)
  Vdss | 6710 (1700)

18. Secondary Outcome: Total Body Effective Half-life (EHL)
Description: Total body EHL is the time required for a radioactive element in the body to be diminished by 50% as a result of radioactive decay and biologic elimination. The EHL is equal to the product of the biologic half-life (BHL) and the radioactive half-life (RHL) divided by the sum of the BHL and the RHL: EHL=(BHL * RHL)/(BHL + RHL). BHL is the time it takes for a drug to lose half of its pharmacologic, physiologic, or radiologic activity. RHL is the time taken for half of the radioactive nuclei to decay.
Time Frame: as for outcome 12
Population: ITT-Exposed Population
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Tositumomab and Iodine I-131 Tositumomab
Number analyzed (Participants) | 76
hours | 63.6 (8.44)

19. Secondary Outcome: Normal Organ Dosimetry for the Indicated Organs
Description: Organ dosimetry was performed in participants using the kidneys, liver, lungs, spleen, red marrow, urinary bladder, and the remainder of the body as source organs. Organ doses and Iodine I-131 Anti-B1 Antibody biodistribution were comparable across the three Anti-B1 Antibody manufacturers. Gamma camera images of participants were used to calculate the amount of radiation that accumulated in the target tumor and normal organs (tumor/organ dosimetry). For the spleen (corrected) category, participant-specific corrections were made to account for individual spleen size.
Time Frame: as for outcome 12
Population: ITT-Exposed Population. Only those participants who had available gamma camera images for the indicated organs were assessed.
Measure: Mean (Standard Deviation); unit: cGy/75 cGy total body dose (TBD)
Arm/Group | Tositumomab and Iodine I-131 Tositumomab
Number analyzed (Participants) | 76
cGy/75 cGy total body dose (TBD)
  Liver, n=76 | 221.69 (43.721)
  Kidney, n=75 | 637.35 (129.360)
  Spleen, n=74 | 835.92 (358.610)
  Spleen (corrected), n=72 | 393.38 (120.602)
  Blood, n=76 | 364.60 (64.608)
  Red Bone Marrow, n=41 | 105.57 (10.342)
  Thyroid, n=76 | 59.50 (3.170)
  Urine Bladder Wall, n=76 | 214.28 (38.563)
  Gall Bladder Wall, n=76 | 89.39 (3.929)
  Tumor, n=61 | 835.86 (499.817)

20. Secondary Outcome: Number of Participants With the Indicated Fatal Serious Adverse Events (SAE)
Description: An SAE is any event occurring at any dose that results in any of the following: death, a life-threatening adverse drug experience (ADE; at immediate risk of death from the experience as it occurred), inpatient hospitalization/prolongation of existing hospitalization, a persistent/significant disability/incapacity, or a congenital anomaly/birth defect. A fatal SAE is a medical event that results in death.
Time Frame: From Baseline up to 12 years from the start of treatment (long-term follow up)
Population: ITT-Exposed Population
Measure: Number; unit: participants
Arm/Group | Tositumomab and Iodine I-131 Tositumomab
Number analyzed (Participants) | 76
participants | 1

21. Secondary Outcome: Number of Participants Evaluable and Not Evaluable for Human Anti-Murine Antibodies (HAMA)
Description: Tositumomab is a murine (mouse) antibody (immunoglobulin) of the IgG2a subclass. Participants were evaluated to determine whether they developed an immune response to study treatment, as evident by human anti-mouse antibodies (HAMA) after administration of tositumomab and iodine I-131 tositumomab. A positive HAMA value indicates that the participant developed HAMA above the HAMA assay threshold, and a negative HAMA value indicates either the absence or below threshold level of HAMA.
Time Frame: From Baseline up to 2 years from the start of treatment
Population: ITT-Exposed Population
Measure: Number; unit: participants
Arm/Group | Tositumomab and Iodine I-131 Tositumomab
Number analyzed (Participants) | 76
participants
  Evaluable | 73
  Not evaluable | 3

22. Secondary Outcome: Number of Participants With Conversion to HAMA Positivity Any Time During the Study From Baseline
Description: Tositumomab is a murine (mouse) antibody (immunoglobulin) of the IgG2a subclass. Participants were evaluated to determine whether they developed an immune response to study treatment, as evident by human anti-mouse antibodies (HAMA) after administration of tositumomab and iodine I-131 tositumomab. A positive HAMA value indicates that the participant developed HAMA above the HAMA assay threshold, and a negative HAMA value indicates either the absence or below threshold level of HAMA. HAMA assays were conducted in the laboratory to measure conversion to HAMA positivity following treatment.
Time Frame: From Baseline up to 2 years from the start of treatment
Population: ITT-Exposed Population. Only those participants who were evaluable for HAMA were assessed.
Measure: Number; unit: participants
Arm/Group | Tositumomab and Iodine I-131 Tositumomab
Number analyzed (Participants) | 73
participants
  Positive | 51
  Negative | 22

23. Secondary Outcome: Time to HAMA Positivity From the First Dosimetric Dose
Description: as for outcome 22
Time Frame: From Baseline up to 2 years from the start of treatment
Population: ITT-Exposed Population. Only those participants who converted from being negative for HAMA at Baseline to being positive for HAMA any time following treatment were assessed.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Tositumomab and Iodine I-131 Tositumomab
Number analyzed (Participants) | 51
days | 93.5 (152.6)

24. Secondary Outcome: Number of Participants With Elevated, Low, and Normal Thyroid Stimulating Hormone (TSH) Levels at Baseline
Description: TSH is a hormone that stimulates the thyroid gland to produce thyroxine (T4) and then triiodothyronine (T3), which stimulates the metabolism of almost every tissue in the body. Participants were considered to have normal, high, or low TSH levels per the standard TSH ranges of the testing laboratory.
Time Frame: Baseline
Population: ITT-Exposed Population. Only those participants for whom TSH levels were recorded at Baseline were assessed.
Measure: Number; unit: participants
Arm/Group | Tositumomab and Iodine I-131 Tositumomab
Number analyzed (Participants) | 73
participants
  Elevated TSH at Baseline | 4
  Low/Normal TSH at Baseline | 69

25. Secondary Outcome: Participants With Elevated TSH Levels at Baseline With Post Baseline TSH Levels of Low/Normal and Elevated
Description: as for outcome 24
Time Frame: Baseline and up to 12 years (long-term follow up)
Population: ITT-Exposed Population. Only participants with elevated TSH levels at Baseline were assessed.
Measure: Number; unit: participants
Arm/Group | Tositumomab and Iodine I-131 Tositumomab
Number analyzed (Participants) | 73
participants
  Low/Normal TSH Post Baseline | 61
  Elevated TSH Post Baseline | 8

26. Secondary Outcome: Time to Elevated TSH Post Baseline for Participants Who Had Low or Normal TSH Levels at Baseline and Elevated Levels Post Baseline
Description: TSH is a hormone that stimulates the thyroid gland to produce thyroxine (T4) and then triiodothyronine (T3), which stimulates the metabolism of almost every tissue in the body. Participants were categorized to have elevated or normal/low TSH values per the standard TSH ranges of the testing laboratory.
Time Frame: Baseline and up to 12 years from the start of treatment
Population: ITT-Exposed Population. Only those participants who had low or normal TSH levels at Baseline and elevated levels post Baseline were assessed.
Measure: Median (Full Range); unit: months
Arm/Group | Tositumomab and Iodine I-131 Tositumomab
Number analyzed (Participants) | 8
months | 33.2 [5.9 to 106.2]

27. Secondary Outcome: Number of Participants With the Adverse Event (AEs) of Hypothyroidism
Description: Hypothyroidism is a condition in which the thyroid gland does not make enough thyroid hormone and is defined as either developing elevated TSH levels or initiating thyroid medication. An AE is defined as any unfavorable and unintended sign, including an abnormal laboratory finding, symptom, or disease associated with the use of a medical treatment or procedure, regardless of whether it is considered to be related to the medical treatment or procedure, that occurs during the course of the study.
Time Frame: Baseline and up to 12 years from the start of treatment
Population: ITT-Exposed Population
Measure: Number; unit: participants
Arm/Group | Tositumomab and Iodine I-131 Tositumomab
Number analyzed (Participants) | 76
participants | 8

28. Secondary Outcome: Number of Participants With Low or Normal Baseline TSH Levels That Developed Hypothyroidism
Description: Hypothyroidism is a condition in which the thyroid gland does not make enough thyroid hormone and is defined as either developing elevated TSH levels or initiating thyroid medication.
Time Frame: Baseline and up to 12 years from the start of treatment
Population: ITT-Exposed Population. Only those participants who had low or normal Baseline TSH levels were assessed.
Measure: Number; unit: participants
Arm/Group | Tositumomab and Iodine I-131 Tositumomab
Number analyzed (Participants) | 69
participants | 6

29. Secondary Outcome: Number of Participants Who Received Thyroid Medication After Treatment
Description: as for outcome 28
Time Frame: From Study Day 0 (start of treatment) up to 12 years (long-term follow up)
Population: ITT-Exposed Population
Measure: Number; unit: participants
Arm/Group | Tositumomab and Iodine I-131 Tositumomab
Number analyzed (Participants) | 76
participants | 11

ADVERSE EVENTS:
Time Frame: Serious adverse events (SAEs) and non-serious AEs were collected from Baseline (Study Day 0) until 12 years follow-up from the start of treatment.
Arm/Group | Tositumomab and Iodine I-131 Tositumomab
Serious Adverse Events (participants affected / at risk) | 19/76
Other Adverse Events (participants affected / at risk) | 76/76
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tositumomab and Iodine I-131 Tositumomab (N=76)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Breast cancer in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Endometrial cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Glioblastoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Hyperthyroidism (Endocrine disorders) | 1
Hypothyroidism (Endocrine disorders) | 1
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 2
Abdominal pain (Gastrointestinal disorders) | 1
Chest pain (General disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tositumomab and Iodine I-131 Tositumomab (N=76)
Fatigue (General disorders) | 41
Pyrexia (General disorders) | 36
Chills (General disorders) | 19
Oedema peripheral (General disorders) | 9
Feeling cold (General disorders) | 4
Influenza like illness (General disorders) | 4
Local swelling (General disorders) | 4
Pain (General disorders) | 4
Axillary pain (General disorders) | 3
Feeling hot (General disorders) | 3
Malaise (General disorders) | 3
Chest discomfort (General disorders) | 2
Swelling (General disorders) | 2
Asthenia (General disorders) | 1
Catheter site pain (General disorders) | 1
Chest pain (General disorders) | 1
Discomfort (General disorders) | 1
Facial pain (General disorders) | 1
Gait disturbance (General disorders) | 1
Injection site irritation (General disorders) | 1
Sensation of pressure (General disorders) | 1
Nausea (Gastrointestinal disorders) | 52
Vomiting (Gastrointestinal disorders) | 15
Diarrhoea (Gastrointestinal disorders) | 13
Constipation (Gastrointestinal disorders) | 8
Dyspepsia (Gastrointestinal disorders) | 6
Abdominal pain (Gastrointestinal disorders) | 5
Abdominal pain upper (Gastrointestinal disorders) | 5
Abdominal discomfort (Gastrointestinal disorders) | 4
Dysphagia (Gastrointestinal disorders) | 3
Flatulence (Gastrointestinal disorders) | 3
Abdominal distension (Gastrointestinal disorders) | 2
Gastritis (Gastrointestinal disorders) | 2
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 2
Mouth ulceration (Gastrointestinal disorders) | 2
Aphthous stomatitis (Gastrointestinal disorders) | 1
Cheilitis (Gastrointestinal disorders) | 1
Dry mouth (Gastrointestinal disorders) | 1
Faecal incontinence (Gastrointestinal disorders) | 1
Glossodynia (Gastrointestinal disorders) | 1
Haematemesis (Gastrointestinal disorders) | 1
Hypoaesthesia oral (Gastrointestinal disorders) | 1
Lip swelling (Gastrointestinal disorders) | 1
Oral disorder (Gastrointestinal disorders) | 1
Stomatitis (Gastrointestinal disorders) | 1
Swollen tongue (Gastrointestinal disorders) | 1
Tooth disorder (Gastrointestinal disorders) | 1
Toothache (Gastrointestinal disorders) | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 34
Arthralgia (Musculoskeletal and connective tissue disorders) | 33
Neck pain (Musculoskeletal and connective tissue disorders) | 10
Back pain (Musculoskeletal and connective tissue disorders) | 9
Pain in extremity (Musculoskeletal and connective tissue disorders) | 9
Joint swelling (Musculoskeletal and connective tissue disorders) | 7
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 6
Muscle spasms (Musculoskeletal and connective tissue disorders) | 3
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 3
Joint stiffness (Musculoskeletal and connective tissue disorders) | 2
Muscular weakness (Musculoskeletal and connective tissue disorders) | 2
Pain in jaw (Musculoskeletal and connective tissue disorders) | 2
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 1
Headache (Nervous system disorders) | 42
Dizziness (Nervous system disorders) | 10
Dysgeusia (Nervous system disorders) | 5
Paraesthesia (Nervous system disorders) | 3
Hypoaesthesia (Nervous system disorders) | 2
Somnolence (Nervous system disorders) | 2
Hyperaesthesia (Nervous system disorders) | 1
Lethargy (Nervous system disorders) | 1
Memory impairment (Nervous system disorders) | 1
Migraine (Nervous system disorders) | 1
Poor quality sleep (Nervous system disorders) | 1
Sensory disturbance (Nervous system disorders) | 1
Sinus headache (Nervous system disorders) | 1
Syncope (Nervous system disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 28
Rash (Skin and subcutaneous tissue disorders) | 13
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 12
Rash generalised (Skin and subcutaneous tissue disorders) | 7
Urticaria (Skin and subcutaneous tissue disorders) | 7
Rash pruritic (Skin and subcutaneous tissue disorders) | 6
Erythema (Skin and subcutaneous tissue disorders) | 4
Night sweats (Skin and subcutaneous tissue disorders) | 3
Swelling face (Skin and subcutaneous tissue disorders) | 3
Alopecia (Skin and subcutaneous tissue disorders) | 2
Rash erythematous (Skin and subcutaneous tissue disorders) | 2
Circumoral oedema (Skin and subcutaneous tissue disorders) | 1
Ecchymosis (Skin and subcutaneous tissue disorders) | 1
Exfoliative rash (Skin and subcutaneous tissue disorders) | 1
Pain of skin (Skin and subcutaneous tissue disorders) | 1
Palmar erythema (Skin and subcutaneous tissue disorders) | 1
Petechiae (Skin and subcutaneous tissue disorders) | 1
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 1
Pruritus generalised (Skin and subcutaneous tissue disorders) | 1
Rash papular (Skin and subcutaneous tissue disorders) | 1
Skin burning sensation (Skin and subcutaneous tissue disorders) | 1
Skin discolouration (Skin and subcutaneous tissue disorders) | 1
Skin lesion (Skin and subcutaneous tissue disorders) | 1
Skin odour abnormal (Skin and subcutaneous tissue disorders) | 1
Telangiectasia (Skin and subcutaneous tissue disorders) | 1
Decreased appetite (Metabolism and nutrition disorders) | 40
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 12
Cough (Respiratory, thoracic and mediastinal disorders) | 6
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 6
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 6
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 3
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 3
Nasal discomfort (Respiratory, thoracic and mediastinal disorders) | 2
Productive cough (Respiratory, thoracic and mediastinal disorders) | 2
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 2
Sneezing (Respiratory, thoracic and mediastinal disorders) | 2
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1
Pharyngeal oedema (Respiratory, thoracic and mediastinal disorders) | 1
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1
Throat tightness (Respiratory, thoracic and mediastinal disorders) | 1
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1
White Blood Cells (WBC) < 2000 cells/cubic millimeter (CMM) (Investigations) | 22
Absolute neutrophil count (ANC) < 1000 Cells/CMM (Investigations) | 20
Platelets < 50000 cells/CMM (Investigations) | 13
Upper respiratory tract infection (Infections and infestations) | 8
Nasopharyngitis (Infections and infestations) | 4
Sinusitis (Infections and infestations) | 3
Diarrhoea infectious (Infections and infestations) | 1
Folliculitis (Infections and infestations) | 1
Fungal infection (Infections and infestations) | 1
Gastroenteritis viral (Infections and infestations) | 1
Herpes simplex (Infections and infestations) | 1
Herpes zoster (Infections and infestations) | 1
Influenza (Infections and infestations) | 1
Laryngitis (Infections and infestations) | 1
Oral herpes (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 1
Rash pustular (Infections and infestations) | 1
Respiratory tract infection viral (Infections and infestations) | 1
Rhinitis (Infections and infestations) | 1
Insomnia (Psychiatric disorders) | 12
Anxiety (Psychiatric disorders) | 8
Depression (Psychiatric disorders) | 3
Agitation (Psychiatric disorders) | 1
Depressed mood (Psychiatric disorders) | 1
Emotional poverty (Psychiatric disorders) | 1
Hallucination (Psychiatric disorders) | 1
Nightmare (Psychiatric disorders) | 1
Flushing (Vascular disorders) | 10
Hot flush (Vascular disorders) | 2
Hypotension (Vascular disorders) | 2
Hypertension (Vascular disorders) | 1
Peripheral coldness (Vascular disorders) | 1
Lymphadenopathy (Blood and lymphatic system disorders) | 8
Lymph node pain (Blood and lymphatic system disorders) | 6
Conjunctivitis (Eye disorders) | 7
Eye irritation (Eye disorders) | 2
Lacrimation increased (Eye disorders) | 2
Ocular hyperaemia (Eye disorders) | 2
Photophobia (Eye disorders) | 2
Vision blurred (Eye disorders) | 2
Conjunctival hyperaemia (Eye disorders) | 1
Eye oedema (Eye disorders) | 1
Eye pain (Eye disorders) | 1
Eye pruritus (Eye disorders) | 1
Eye swelling (Eye disorders) | 1
Eyelid oedema (Eye disorders) | 1
Body temperature increased (Investigations) | 6
Blood pressure decreased (Investigations) | 1
Blood thyroid stimulating hormone increased (Investigations) | 1
Electrocardiogram abnormal (Investigations) | 1
Weight decreased (Investigations) | 1
Weight increased (Investigations) | 1
Menstruation irregular (Reproductive system and breast disorders) | 5
Amenorrhoea (Reproductive system and breast disorders) | 2
Breast tenderness (Reproductive system and breast disorders) | 1
Menopausal symptoms (Reproductive system and breast disorders) | 1
Pelvic pain (Reproductive system and breast disorders) | 1
Vaginal haemorrhage (Reproductive system and breast disorders) | 1
Hypothyroidism (Endocrine disorders) | 7
Hyperthyroidism (Endocrine disorders) | 1
Ear pruritus (Ear and labyrinth disorders) | 5
Ear congestion (Ear and labyrinth disorders) | 1
Ear discomfort (Ear and labyrinth disorders) | 1
Procedural pain (Injury, poisoning and procedural complications) | 2
Contusion (Injury, poisoning and procedural complications) | 1
Forearm fracture (Injury, poisoning and procedural complications) | 1
Post procedural discomfort (Injury, poisoning and procedural complications) | 1
Wound (Injury, poisoning and procedural complications) | 1
Tachycardia (Cardiac disorders) | 2
Aortic valve incompetence (Cardiac disorders) | 1
Atrioventricular block (Cardiac disorders) | 1
Mitral valve incompetence (Cardiac disorders) | 1
Palpitations (Cardiac disorders) | 1
Pericardial effusion (Cardiac disorders) | 1
Tricuspid valve incompetence (Cardiac disorders) | 1
Ventricular tachycardia (Cardiac disorders) | 1
Chromaturia (Renal and urinary disorders) | 1
Nocturia (Renal and urinary disorders) | 1
Urinary incontinence (Renal and urinary disorders) | 1
Urine odour abnormal (Renal and urinary disorders) | 1
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.